CLINICAL TRIAL: NCT03530644
Title: Comparative Study Between Two Models of a Non-invasive Glucose Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RSP-14
Record Dates: First submitted 2018-04-11; First posted 2018-05-21 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Type1diabetes
Keywords: Non-invasive glucose monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSP-14 (Experimental): Comparative study of two Investigational Medical Devices (WM3.4NR and P0.1)
  Optical data will be obtained from T1D over a dynamic glycemic range. Data will be paired with references.
  Interventions: Device: WM3.4NR; Device: P0.1

INTERVENTIONS:
Device: WM3.4NR — The investigational medical device will collect spectral Raman data from tissue.
Device: P0.1 — The investigational medical device will collect spectral Raman data from tissue.

SUMMARY:
This clinical study has been launched to compare the performances of two models of a non-invasive glucose monitoring device.

DETAILED DESCRIPTION:
Subjects will be optical screened at baseline visit. Study comprises two in-clinic visits. Subjects will arrive in a fasting state and and oral glucose bolus will be administered.

Subjects will during each of two study days be subjected to optical readings on two different device prototypes. During each of the study days, FGM readings, capillary blood samples and arterialized venous blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older
* Diabetic type 1 patients
* Insulin pump users
* Skin phototype 1-4

Exclusion Criteria:

* For female participants: Pregnancy or subject is attempting to conceive or not willing and able to practice birth control during the study duration
* For female participants: Breastfeeding
* Subjects not able to understand and read Danish
* In Investigator's opinion, subject is not able to follow instructions as specified in the protocol
* Rejection by optical screenings
* Subjects not able to hold hand/arm steadily (including tremors and Parkinson's Disease)
* Diagnosed with reduced circulation
* Extensive skin changes, tattoos or diseases on probe application site
* Known allergy to medical grade alcohol
* Known allergy to adhesives
* Systemic or topical administration of glucocorticoids for the past 7 days
* Subjects undergoing dialysis treatment
* Medical history or any condition that may, in the opinion of the Investigator, compromise the subject's ability to participate
* Concomitant medical condition which could present a risk to the safety or welfare of the subject or study staff
* Subjects currently enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Generation and validation of prediction models | 4 months
  Two in-clinic visits each of a duration of 7-8 hours are scheduled for each subject. Subjects will enter clinic in fasting state and will receive an oral glucose bolus. Glucose excursion is followed with frequent capillary and venous blood samples along with FGM readings. In parallel, optical glucose data from two different prototypes of the investigational medical device will be collected.
  Optical glucose readings will be masked to the subjects.
  Collected data will be used to generate individual calibration models capable of predicting tissue glucose. Models from the two devices will be validated on independent data sets using MARD, ISUP and Consensus Error Grid endpoint measures.
Performance evaluation | 4 months
  Validated calibration models will be compared with MARD, ISUP and Consensus Error Grid endpoint measures.

SECONDARY OUTCOMES:
Safety by paucity of adverse events | 4 months
  To evaluate safety of devices in a descriptive manner by the paucity of adverse events. Adverse events will be recorded during study.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, PhD, Principal Investigator — Steno Diabetes Center Odense, Denmark; Vibe Vestergaard, Nurse, Principal Investigator — Steno Diabetes Center Odense, Denmark
Locations (1):
- Steno Diabetes Center Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No